CLINICAL TRIAL: NCT00029224
Title: A Prospective, Multicenter, Open-label Clinical Evaluation of the Effect of IV Zoledronic Acid 4mg on PAIN, QUALITY OF LIFE and TIME IN INFUSION CHAIR in Breast Cancer, Multiple Myeloma, and Prostate Cancer Patients With Cancer-related Bone Lesions
Brief Title: Treatment With Zoledronic Acid in Patients With Breast Cancer, Multiple Myeloma, and Prostate Cancer With Cancer Related Bone Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EUS16
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer; Multiple Myeloma; Prostate Cancer
Keywords: bone lesions; breast cancer; multiple myeloma; prostate cancer; bone metastases; pain
MeSH Terms: conditions — Breast Neoplasms; Multiple Myeloma; Prostatic Neoplasms; Pain | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
Patients with bone metastases or bone lesions caused by breast cancer, multiple myeloma or prostate cancer will be treated with IV Zometa in a 15 minute infusion. Pain will be evaluated, as well as time in chair, quality of life and safety of Zometa.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent
* Greater than 18 years of age
* Proof of breast cancer, multiple myeloma or prostate cancer
* Diagnosis of at least one cancer-related bone lesion
* If patient is of child-bearing potential, negative pregnancy test and on a medically recognized form of contraception
* ECOG performance status of 0,1 or 2
* Ability to read, understand and write English or Spanish language
* Normal renal function
* Corrected serum calcium equal to or greater than 8mg/dl Exclusion Criteria
* clinically symptomatic brain metastases
* hypersensitivity to Zometa or other bisphosphonates
* pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2001-10; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Pain score assessed by change from baseline

SECONDARY OUTCOMES:
Quality of life
Time in infusion chair
Safety assessed by adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - Osceola Cancer Center, Kissimmee, Florida
  - Nevada Cancer Center, Las Vegas, Nevada
  - Hematology-Oncology Associates PC, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Medforo, Oregon
  - Virginia Physicians, Inc, Richmond, Virginia